CLINICAL TRIAL: NCT04613375
Title: Low Intervention Study of the Effectiveness Of 13-Valent Pneumococcal Conjugate Vaccine (PCV13) Against Vaccine Type Pneumococcal Hospitalised Community Acquired Pneumonia (CAP) in Adults 60 Years and Older Using A Test Negative Design Study in A Well-Defined Area of the South of Madrid Region
Brief Title: PCV13 Effectiveness Study Against Hospitalised VT Pneumococcal CAP in Adults 60 Years and Older
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851202; CIBELES (Other: Alias Study Number)
Record Dates: First submitted 2020-10-19; First posted 2020-11-03 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Community Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants
  Interventions: Diagnostic Test: Urine sample collection; Diagnostic Test: Saliva collection

INTERVENTIONS:
Diagnostic Test: Urine sample collection — Serotype specific UAD (urinary antigen detection) test
Diagnostic Test: Saliva collection — Streptococcus pneumonia identification in saliva samples by culture or PCR / RSV identification in saliva samples by PCR

SUMMARY:
Low interventional, prospective, multicentre, hospital-based study involving adults 60 years of age and older hospitalised with CAP at participating sites.

DETAILED DESCRIPTION:
PCV13 efficacy for the prevention of vaccine-type community-acquired pneumonia (VT-CAP) and invasive pneumococcal disease (IPD) was established in the Community-acquired Pneumonia Immunization Trial in Adults (CAPITA) aged 65 and older. However, there are still few available real-life effectiveness estimates in adults. The aim of this study is to evaluate the PCV13 vaccine effectiveness (VE) against hospitalised VT-pneumococcal CAP among adults aged ≥60 years in the Region of Madrid (Spain). Determination of the effectiveness of PCV13 to prevent hospitalised vaccine-type (VT)-pneumococcal CAP among adults aged ≥60 years in Madrid will be evaluated using a test-negative design study, overall and among immunocompetent persons only.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years.
2. Evidence of pneumonia within first 48 hours of hospital admission
3. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Any patient who develops signs and symptoms of pneumonia after being hospitalized for ≥48 hours (either at current hospital, another transferring hospital, or a combination of these).
2. Previously enrolled subjects readmitted ≤14 days after discharge for their study qualifying admission.
3. At the time of enrollment, pneumonia has been excluded as the diagnosis or another diagnosis confirmed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, aged 60 years and over, who are hospitalized with CAP in one of the study hospitals: Hospital Universitario de Móstoles, Hospital Universitario Fundación de Alcorcón, and Hospital Rey Juan Carlos de Móstoles.
Sampling Method: Non-Probability Sample
Enrollment: 1821 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2024-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Spain (5):
  - Hospital Universitarios De Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón
  - Hospital Universitario Rey Juan carlos, Móstoles
  - Hospital Universitario de Mostoles, Móstoles

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851202

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were evaluated for effectiveness of 13-valent pneumococcal conjugate vaccine (PCV13) [received previously at least 30 days before hospitalization] in preventing vaccine-type (VT) pneumococcal hospitalized community acquired pneumonia (CAP) among adults aged greater than or equal to (>=) 60 years in Madrid in this observational study.
Pre-assignment Details: A total of 1821 participants were enrolled in this study and 51 participants did not meet inclusion/exclusion of the study. In this study, a) pandemic period included data from 12 March 2021 to 31 July 2022 when last relevant coronavirus disease 2019 (COVID-19) wave in target population (aged >=60 years) ended in Madrid; b) post-pandemic period included data from 01 August 2022 to 13 September 2023.
Groups:
- All Participants: Eligible participants who were hospitalized with CAP in one of the study hospitals, their data were observed for effectiveness of PCV13 (received previously, not in this study) in this observational study.
Period: Overall Study
Arm/Group | All Participants
Started (Enrolled Population) | 1821
Per-protocol Population | 1770
CAP Population | 1680
CAP Urinary Antigen Detection (UAD) Population | 1512
Completed | 1620
Not Completed | 201
Not completed — Death | 198
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: The per-protocol population included all participants in all enrolled population who met all inclusion/exclusion criteria.
Arm/Group | All Participants
Number analyzed (Participants) | 1770
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.08 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 761
  Male | 1009
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized as Cases and Controls to Determine Vaccine Effectiveness (VE) of PCV13 Against Hospitalized VT CAP: Overall
Description: Cases were participants with CAP with a valid urinary antigen detection (UAD) result in whom PCV13 serotypes were identified by any method. Controls were participants with CAP with a valid UAD result and without having PCV13 serotype. VE was calculated as 1 minus the odd ratio comparing the odds of having received PCV13 for cases and controls, multiplied by 100%. VE is reported as part of statistical data in this outcome measure.
Time Frame: Approximately 30 months
Population: CAP UAD population included all enrolled population who met all inclusion/exclusion criteria and who had a final diagnosis consistent with CAP with a valid UAD result.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 1512
Participants
  Cases | 105
  Controls | 1407
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.3685, Wald Test; Adjusted VE = 16.91, 95% CI 2-sided [-24.43 to 44.52] — Adjusted for the covariates age group, weekly exposure to children less than 5 years, calendar time, and CAP with respiratory syncytial virus (RSV) infection

2. Secondary Outcome: Number of Participants Categorized as Cases and Controls to Determine Vaccine Effectiveness (VE) of PCV13 Against Hospitalized VT CAP By Time Since Vaccination: Overall
Description: Cases were participants with CAP with a valid UAD result in whom PCV13 serotypes were identified by any method. Controls were participants with CAP with a valid UAD result and without having PCV13 serotype. VE was calculated as 1 minus the odd ratio comparing the odds of having received PCV13 for cases and controls, multiplied by 100%. Data is presented in this outcome by time since vaccination. VE is reported as part of statistical data in this outcome measure.
Time Frame: Approximately 30 months
Population: CAP UAD population included all enrolled population who met all inclusion/exclusion criteria and who had a final diagnosis consistent with CAP with a valid UAD result. Here, "Number Analyzed" signifies participants who were evaluable for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 1501
Participants
  Received PCV13 in <2 years or not received PCV13: number analyzed (Participants) | 976
  Received PCV13 in <2 years or not received PCV13: Cases | 66
  Received PCV13 in <2 years or not received PCV13: Controls | 910
  Received PCV13 in 2-<5 years or not received PCV13: number analyzed (Participants) | 1205
  Received PCV13 in 2-<5 years or not received PCV13: Cases | 89
  Received PCV13 in 2-<5 years or not received PCV13: Controls | 1116
  Received PCV13 in >=5 years or not received PCV13: number analyzed (Participants) | 899
  Received PCV13 in >=5 years or not received PCV13: Cases | 66
  Received PCV13 in >=5 years or not received PCV13: Controls | 833
Statistical Analysis 1: Comparison: All Participants; <2 years; Test type: Other; p = 0.0817, Wald Test; Adjusted VE = 49.27, 95% CI 2-sided [-8.9 to 76.37] — Adjusted for the covariates age group, weekly exposure to children less than 5 years, calendar time, and CAP with RSV infection
Statistical Analysis 2: Comparison: All Participants; 2 years to <5 years; Test type: Other; p = 0.8367, Wald Test; Adjusted VE = 4.72, 95% CI 2-sided [-50.96 to 39.87] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: All Participants; >=5 years; Test type: Other; p = 0.7469, Wald Test; Adjusted VE = 12.02, 95% CI 2-sided [-91.53 to 59.59] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of CAP Participants Categorized Per Pneumococcal Serotypes Identified
Description: Percentage of CAP participants in whom streptococcus pneumoniae was identified for PCV13 and 20-valent pneumococcal conjugate vaccine (PCV20) serotypes is reported.
Time Frame: Approximately 30 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of CAP participants
Arm/Group | All Participants
Number analyzed (Participants) | 1512
Percentage of CAP participants
  PCV13 Serotypes | 6.9 [5.7 to 8.3]
  PCV20 Serotypes | 13.2 [11.5 to 15.0]

4. Secondary Outcome: Percentage of CAP Participants in Whom Pneumococcus Identified From Saliva by Culture or Polymerase Chain Reaction (PCR)
Description: Respiratory pneumococcal carriage was determined by testing saliva specimens using both conventional culture and the sensitive molecular method of PCR for the detection of two target genes (lytA and piaB).
Time Frame: Approximately 30 months
Population: CAP UAD population included all enrolled population who met all inclusion/exclusion criteria and who had a final diagnosis consistent with CAP with a valid UAD result. Here, "Number of Participants Analyzed" signifies participants who had a valid saliva specimen test result.
Measure: Number (95% Confidence Interval); unit: Percentage of CAP participants
Arm/Group | All Participants
Number analyzed (Participants) | 1314
Percentage of CAP participants | 11.6 [9.9 to 13.4]

5. Secondary Outcome: Percentage of CAP Participants With Underlying At-risk Medical Conditions
Description: At-risk medical conditions included: alcoholism, asthma, celiac disease, chronic liver disease with hepatic failure, chronic liver disease without hepatic failure, chronic neurologic diseases, chronic obstructive pulmonary disease, coagulation factor replacement therapy, cochlear implant, congestive heart failure, coronary artery disease, cerebrospinal fluid leak, diabetes treated with medication, down syndrome, living in a nursing home, living in a long-term care facility, occupational risk with exposure to metal fumes, other chronic heart disease, other chronic lung disease, other pneumococcal disease risk factors, previous invasive pneumococcal disease, tobacco smoking (tobacco/e-cigarettes).
Time Frame: Approximately 30 months
Population: as for outcome 1
Measure: Number; unit: Percentage of CAP participants
Arm/Group | All Participants
Number analyzed (Participants) | 1512
Percentage of CAP participants | 55.2

6. Secondary Outcome: Percentage of CAP Participants With Underlying at High-Risk Medical Conditions
Description: High-risk medical conditions included: asplenia, cancer/malignancy (hematologic), cancer/malignancy (solid tumor), chronic kidney disease, human immunodeficiency virus (HIV) - acquired immunodeficiency syndrome (AIDS), HIV - No AIDS, immunodeficiency, immunosuppressant drug therapy, multiple myeloma, organ transplantation.
Time Frame: Approximately 30 months
Population: as for outcome 1
Measure: Number; unit: Percentage of CAP participants
Arm/Group | All Participants
Number analyzed (Participants) | 1512
Percentage of CAP participants | 35.6

7. Secondary Outcome: Percentage of Streptococcus Pneumoniae (SP) Isolates With Antibiotic Resistance
Description: Percentage of SP isolates with antibiotic resistance to penicillin, amoxicillin, cefotaxime, erythromycin, tetracycline, levofloxacin were reported in this outcome measure.
Time Frame: Approximately 30 months
Population: CAP UAD population included all enrolled population who met all inclusion/exclusion criteria and who had a final diagnosis consistent with CAP with a valid UAD result. Here, "Number of Participants Analyzed" = participants in CAP UAD population from whom valid SP isolates were obtained; "Number of SP isolates analyzed" = number of SP isolates with antimicrobial susceptibility tests performed. Only isolates with antimicrobial susceptibility tests performed were included in analysis.
Measure: Number; unit: Percentage of SP isolates
Units Other Than Participants: SP isolates
Arm/Group | All Participants
Number analyzed (Participants) | 33
Number analyzed (SP isolates) | 33
Percentage of SP isolates
  Penicillin | 9.1
  Amoxicillin | 9.1
  Cefotaxime | 3.0
  Erythromycin | 12.1
  Tetracycline | 12.1
  Levofloxacin | 3.0

8. Post Hoc Outcome: Number of Participants Categorized as Cases and Controls to Determine VE of PCV13 Against Hospitalized VT CAP: Post-Pandemic Period
Description: Cases were participants with CAP with a valid UAD result in whom PCV13 serotypes were identified by any method. Controls were participants with CAP with a valid UAD result and without having PCV13 serotype. VE was calculated as 1 minus the odd ratio comparing the odds of having received PCV13 for cases and controls, multiplied by 100%. VE is reported as part of statistical data in this outcome measure.
Time Frame: Approximately 13.5 months
Population: CAP UAD population included all enrolled population who met all inclusion/exclusion criteria and who had a final diagnosis consistent with CAP with a valid UAD result. Here, "Number of Participants Analyzed" signifies participants in CAP UAD population for post-pandemic period.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 1241
Participants
  Cases | 89
  Controls | 1152
Statistical Analysis 1: Comparison: All Participants; Test type: Other; p = 0.1827, Wald Test; Adjusted VE = 25.96, 95% CI 2-sided [-15.21 to 52.42] — [estimate comment as in outcome 2, analysis 1]

9. Post Hoc Outcome: Number of Participants Categorized as Cases and Controls to Determine Vaccine Effectiveness (VE) of PCV13 Against Hospitalized VT CAP By Time Since Vaccination: Post-pandemic Period
Description: as for outcome 2
Time Frame: Approximately 13.5 months
Population: CAP UAD population included all enrolled population who met all inclusion/exclusion criteria and who had a final diagnosis consistent with CAP with a valid UAD result. Here, "Number of Participants Analyzed" signifies participants in CAP UAD population for post-pandemic period and "Number Analyzed" signifies participants who were evaluable for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 1241
Participants
  Received PCV13 in <2 years or not received PCV13: number analyzed (Participants) | 778
  Received PCV13 in <2 years or not received PCV13: Cases | 55
  Received PCV13 in <2 years or not received PCV13: Controls | 723
  Received PCV13 in 2-<5 years or not received PCV13: number analyzed (Participants) | 999
  Received PCV13 in 2-<5 years or not received PCV13: Cases | 79
  Received PCV13 in 2-<5 years or not received PCV13: Controls | 920
  Received PCV13 in >=5 years or not received PCV13: number analyzed (Participants) | 724
  Received PCV13 in >=5 years or not received PCV13: Cases | 57
  Received PCV13 in >=5 years or not received PCV13: Controls | 667
Statistical Analysis 1: Comparison: All Participants; <2 years; Test type: Other; p = 0.028, Wald Test; Adjusted VE = 68.86, 95% CI 2-sided [11.86 to 89] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: All Participants; 2 years to <5 years; Test type: Other; p = 0.738, Wald Test; Adjusted VE = 7.97, 95% CI 2-sided [-49.73 to 43.43] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: All Participants; >=5 years; Test type: Other; p = 0.4327, Wald Test; Adjusted VE = 30.06, 95% CI 2-sided [-70.86 to 71.37] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Approximately 30 months
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 198/1680
Serious Adverse Events (participants affected / at risk) | 0/1680
Other Adverse Events (participants affected / at risk) | 0/1680

LIMITATIONS AND CAVEATS:
A post-hoc SAP was developed to remove the COVID-19 pandemic period due to changes in healthcare-seeking behavior, hospital admission, vaccination policies, and CAP etiology that could have affected the validity of the overall results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04613375/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04613375/SAP_001.pdf